CLINICAL TRIAL: NCT05861232
Title: THE EFFECT OF INFORMATIVE ANIMATION WATCHING ON ANXIETY AND FEAR DURING INHALATION THERAPY
Brief Title: The Effect of Watching Informative Animation on Fear and Anxiety in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mukader Kaya (Other)
Responsible Party: Sponsor-Investigator, Mukader Kaya, study director, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.0.01.11/285
Record Dates: First submitted 2023-01-11; First posted 2023-05-16 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Inhalation Therapy; Complications

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): informative animation, anxiety and fear
  Interventions: Behavioral: Behavioral
- No Intervention (No Intervention): Control not anxiety and fear

INTERVENTIONS:
Behavioral: Behavioral — fear and anxiety during inhalation therapy
  Arms: Experimental

SUMMARY:
The aim of this project was to determine the effect of showing informative animations to children on anxiety and fear during inhalation therapy. This project is a randomized controlled trial. The population of the study will consist of children aged 7-12 years who apply to the Pediatric Emergency Department of Atatürk University Research Hospital between July 2022 and July 2023. The sample of the study will consist of children and their parents who present to the clinic on the dates determined, who are willing to participate in the study, and meet the inclusion criteria. Probability sampling will be used to select the sample. ''Introductory Information Form'', ''Child Fear Scale'', ''Facial Expression Rating Scale'' and ''Informative Animation'' will be used for data collection.

DETAILED DESCRIPTION:
Type of Study: The study was designed as a randomized controlled experimental study. Place and Time of Research:

The study will be conducted at Atatürk University Research Hospital Pediatric Emergency Department between July 2022 and July 2023.

Population and Sample of the Study: The population of the study will consist of children aged 7-12 years who apply to the Pediatric Emergency Department of Atatürk University Research Hospital between July 2022 and July 2023.

ELIGIBILITY:
Inclusion Criteria:

* The child is 7-12 years of age
* The family's willingness to participate in the study
* The child's willingness to participate in the study
* The child does not have a chronic disease

Exclusion Criteria:

* The child has a chronic illness
* The child has a neurological or mental impairment
* The child is visually impaired

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2023-07-07 (Estimated); Study Completion 2023-07-07 (Estimated)

PRIMARY OUTCOMES:
Child Fear Scale (CFS) | 12 MONTHS
  The Child Fear Scale was developed by McMurty et al. in 2011 to measure fear in children undergoing painful medical procedures. The Child Fear Scale is a 0-4 Likert type scale showing five different faces, ranging from neutral (0 = no concern at all) to fearful (4 = severe anxiety).

SECONDARY OUTCOMES:
Facial Expressions Rating Scale | 12 MONTHS
  This visual facial scale is a practical method to assess the level of anxiety within a situation. There are six facial expressions, ranging from very happy to very unhappy, and children are asked to choose the one that comes closest to how they feel at that moment. The most positive face is scored as '0' and the most negative face is scored as '5'.

CONTACTS AND LOCATIONS:
Overall Officials: Mukader KAYA, graduate student, Principal Investigator — ATATÜRK UNİVERSITY
Locations (1):
- Ataturk University Faculty of Nursing, Erzurum, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
THE ARTICLE IS INTENDED TO BE SHARED AFTER PUBLICATION.